CLINICAL TRIAL: NCT07325643
Title: Effectiveness of a Hydroxyapatite-Containing Toothpaste Versus Mouthwash in Preventing White-Spot Lesions During Fixed-Appliance Orthodontic Treatment: A Randomized Clinical Trial
Brief Title: Effect of Hydroxyapatite Toothpaste and Mouthwash in Preventing White Spot Lesions During Orthodontic Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heba Tahseen Almasri (Other)
Responsible Party: Sponsor-Investigator, Heba Tahseen Almasri, Principal Investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WLS-HA-Ortho-2025
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Prevention of White Spot Lesions in Patients Undergoing Orthodontic Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAp toothpaste + placebo mouth wash (Experimental): HAp toothpaste + placebo mouthwash
  * Arm Description: Participants will brush their teeth three times daily with hydroxyapatite toothpaste and rinse twice daily with a placebo mouthwash.
  Interventions: Dietary Supplement: Hydroxyapatite Toothpaste
- HAp mouthwash + fl toothpaste (Experimental): Fluoride toothpaste + HAp mouthwash
  * Arm Description: Participants will brush their teeth three times daily with fluoride toothpaste and rinse twice daily with HAp mouthwash.
  Interventions: Dietary Supplement: Hydroxyapatite Mouthwash
- Fluoride toothpaste + placebo mouthwash (Placebo Comparator): Fluoride toothpaste + placebo mouthwash
  * Arm Description: Participants will brush their teeth three times daily with fluoride toothpaste and rinse twice daily with a placebo mouthwash.
  Interventions: Other: Fluoride Toothpaste + Placebo Mouthwash

INTERVENTIONS:
Dietary Supplement: Hydroxyapatite Toothpaste — Participants will brush their teeth three times daily with hydroxyapatite-containing toothpaste to evaluate its effect on preventing white spot lesions during orthodontic treatment.
  Arms: HAp toothpaste + placebo mouth wash
Dietary Supplement: Hydroxyapatite Mouthwash — Participants will rinse their mouth twice daily with hydroxyapatite-containing mouthwash to assess its preventive effect on white spot lesions in orthodontic patients.
  Arms: HAp mouthwash + fl toothpaste
Other: Fluoride Toothpaste + Placebo Mouthwash — Participants will brush their teeth three times daily with fluoride toothpaste and rinse twice daily with placebo mouthwash, serving as the control group for comparison with hydroxyapatite interventions.
  Arms: Fluoride toothpaste + placebo mouthwash

SUMMARY:
This study aims to evaluate the effect of hydroxyapatite-containing toothpaste and mouthwash in preventing white spot lesions in patients undergoing orthodontic treatment.

Participants: 75 patients will be divided into three groups:

* Group A: Participants will brush their teeth three times a day using hydroxyapatite toothpaste and rinse twice a day with a placebo mouthwash.
* Group B: Participants will brush their teeth three times a day using fluoride toothpaste and rinse twice a day with hydroxyapatite mouthwash.
* Group C (Control Group): Participants will brush their teeth three times a day using fluoride toothpaste and rinse twice a day with a placebo mouthwash.

Patients will be followed during their orthodontic treatment to assess the development of white spot lesions.

The study is safe and involves no surgical procedures or risky medications, and will be conducted under the supervision of Principal Investigator Heba Masri after obtaining ethical approval.

DETAILED DESCRIPTION:
This randomized, three-group study aims to evaluate the effectiveness of hydroxyapatite in preventing white spot lesions during orthodontic treatment in patients who initially do not have these lesions.

Study Design:

* Total Participants: 75 patients (25 per group)
* Duration: Throughout orthodontic treatment
* Groups:
* Group A: Brush teeth three times daily with hydroxyapatite toothpaste and rinse twice daily with placebo mouthwash.
* Group B: Brush teeth three times daily with fluoride toothpaste and rinse twice daily with hydroxyapatite mouthwash.
* Group C (Control): Brush teeth three times daily with fluoride toothpaste and rinse twice daily with placebo mouthwash.

Outcome Assessments:

All assessments of white-spot lesions will be performed using Diagnodent Pen, Gorlick index (GI), digital photographs, Gingival Bleeding Index (GBI), Plaque Index (PI), and salivary pH measurements.

Ethical Considerations:

* All participants will sign informed consent prior to joining the study.
* The study was approved by the Ethics Committee, College of Dentistry, University of Baghdad.
* This study involves low-risk interventions (toothpaste and mouthwash) and does not use U.S. FDA-regulated drugs or devices.

Study Objective:

* To determine whether hydroxyapatite-containing toothpaste and/or mouthwash is more effective than conventional products in preventing white spot lesions during orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria: All included participants will be drawn from those who will receive comprehensive orthodontic treatment and fulfill the following inclusion criteria:

1. Complete permanent dentition up to the first premolar, with no intended extractions in orthodontic treatment plan.
2. Good overall health.
3. Good oral hygiene: full-mouth plaque score < 20%.
4. No bleeding upon probing after 30 seconds.
5. Discontinuous band of plaque at the gingival margin.
6. Normal stimulated salivary flow rate.
7. Normal buffer capacity (final pH between 6.0 and 7.0) -

Exclusion Criteria:

* 1. History of previous orthodontic treatment. 2. Bleaching or topical fluoridation within the last six months. 3. Severely rotated any of the study teeth (limiting the appearance of facial surfaces).

  4. Visible signs of caries, fluorosis, hypocalcification, or other developmental defects. 5. Restoration on the labial surface of the study teeth. 6. Systemic or endocrine conditions (e.g., cardiac pacemakers, diabetes mellitus).

  7. Craniofacial anomalies and clefts.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Severity of White Spot Lesions assessed by Gorelick Index | Baseline, 1,3 months, and 6 months
  Severity of white spot lesions on labial tooth surfaces assessed using the Gorelick index during orthodontic treatment.
  Time Frame:
  Baseline to 6 months
  Unit of Measure:
  Score
Enamel Demineralization assessed by DIAGNOdent | Baseline, 1,3 months, and 6 months
  Enamel demineralization level measured using DIAGNOdent laser fluorescence device during orthodontic treatment.
  Unit of Measure:
  DIAGNOdent score (laser fluorescence units)

SECONDARY OUTCOMES:
Plaque Index | Baseline, 1, 3 months, 6 months
  Plaque accumulation assessed using a standardized plaque index during orthodontic treatment.
Gingival Bleeding Index | Baseline, 1,3to and 6 months
  Gingival bleeding assessed using a standardized bleeding index during orthodontic treatment.
Salivary pH | Baseline, 1,3 and 6 months
  Salivary pH measured using pH indicator strips during orthodontic treatment. pH value

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad - College of Dentistry / Orthodontic Clinic, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team due to privacy concerns and the sensitive nature of patient information

REFERENCES:
- [Background] Farook, F.F., 2023. The efficacy of manual toothbrushes in patients with fixed orthodontic appliances: a randomized clinical trial. BMC Oral Health, 23(1), p.35 Gorelick, L., Geiger, A.M. & Gwinnett, A.J., 1982. Incidence of white spot formation after bonding and banding. Am J Orthod, 81(2), pp.93-98 Banks, P. & Richmond, S., 1994. Enamel sealants: a clinical evaluation of their value during fixed appliance therapy. Eur J Orthod, 16(1), pp.19-25 Silness, J. & Löe, H., 1964. Periodontal disease in pregnancy. II. Correlation between oral hygiene and periodontal condition. Acta Odontol Scand, 22(1), pp.121-135 Löe, H. & Silness, J., 1963. Periodontal disease in pregnancy. I. Prevalence and severity. Acta Odontol Scand, 21(6), pp.533-551 Du, M., Cheng, N., Tai, B., Jiang, H., Li, J. & Bian, Z., 2011. Randomized controlled trial on fluoride varnish application for treatment of white spot lesion after fixed orthodontic treatment. Clin Oral Investig, 16(2), pp.463-468. https://doi.org/10.1007/s00784-011-0520-4 Gohar, R.A.A.E.G., Ibrahim, S.H. & Safwat, O.M., 2023. Evaluation of the remineralizing effect of biomimetic self-assembling peptides in post-orthodontic white spot lesions compared to fluoride-based delivery systems: randomized controlled trial. Clin Oral Investig, 27(2), pp.613-624. doi:10.1007/s00784-022-04757-7 Campus, G., Cocco, F., Wierichs, R.J., Wolf, T.G., Salerno, C., Arghittu, A., Dettori, M. & Cagetti, M.G., 2024. Effects of Hydroxyapatite-Containing Toothpastes on Some Caries-Related Variables: A Randomised Clinical Trial. Int Dent J, 74(6), pp.754-761. https://doi.org/10.1016/j.identj.2024.01.028 Alkarad, L., Alkhouli, M. & Dashash, M., 2023. Remineralization of teeth with casein phosphopeptide-amorphous calcium phosphate: analysis of salivary pH and the rate of salivary flow. BDJ Open, 9(1), p.16. doi:10.1038/s41405-023-00141-z
- [Background] Paszyńska, E., Górska, R., Kaczmarek, U., et al., 2023. Caries-preventing effect of a hydroxyapatite-toothpaste in adults: A randomized, double-blind, clinical trial. Frontiers in Public Health, 11, p.1199728. https://doi.org/10.3389/fpubh.2023.1199728 BMC Oral Health, 2022. Effects of hydroxyapatite toothpaste on tooth whitening and enamel remineralization: Clinical evaluation. BMC Oral Health, 22, p.345. https://doi.org/10.1186/s12903-022-02266-3 Saliasi, I., Llodra, J.C., Bravo, M., Tramini, P., Dussart, C., Viennot, S. & Carrouel, F., 2018. Effect of a Toothpaste/Mouthwash Containing Carica papaya Leaf Extract on Interdental Gingival Bleeding: A Randomized Controlled Trial. Int J Environ Res Public Health, 15(12), p.2660. https://doi.org/10.3390/ijerph15122660 Araujo, M.W.B., Charles, C.A., Weinstein, R.B., Parikh-Das, A.M., Zhang, J., & Gunsolley, J.C., 2015. Meta-analysis of the effect of an essential oil-containing mouthrinse on gingivitis and plaque. J Am Dent Assoc, 146(8), pp.610-622. https://doi.org/10.1016/j.adaj.2015.05.007 Hoffman, D.A., Clark, A.E., Rody Jr., W.J., McGorray, S.P. & Wheeler, T.T., 2015. A prospective randomized clinical trial into the capacity of a toothpaste containing NovaMin to prevent white spot lesions and gingivitis during orthodontic treatment. Progress in Orthodontics, 16:25
- [Background] Kouskoura, T., Ochsner, T., Verna, C., Pandis, N. & Kanavakis, G., 2022. The effect of orthodontic treatment on facial attractiveness: a systematic review and meta-analysis. European Journal of Orthodontics, 44(6), pp.636-649. doi:10.1093/ejo/cjat064 Kozak, U., Lasota, A. & Chałas, R., 2021. Changes in distribution of dental biofilm after insertion of fixed orthodontic appliances. Journal of Clinical Medicine, 10(23), p.5638. doi:10.3390/jcm10235638 Lopes, P.C. et al., 2024. White Spot Lesions: Diagnosis and Treatment - A Systematic Review. BMC Oral Health, 24(1), pp.1-10. doi:10.1186/s12903-023-03720-6 Choi, A.L., Sun, G., Zhang, Y. & Grandjean, P., 2012. Developmental fluoride neurotoxicity: a systematic review and meta-analysis. Environmental Health Perspectives, 120(10), pp.1362-1368. doi:10.1289/ehp.1104912 Amaechi, B.T., AbdulAzees, P.A., Alshareif, D.O., Shehata, M.A., Lima, P.P.C.S., Abdollahi, A., Samadi Kalkhorani, P. & Evans, V., 2019. Comparative efficacy of a hydroxyapatite and a fluoride toothpaste for prevention and remineralization of dental caries in children. BDJ Open, 5:18
- See also: Systematic review on white spot lesions: diagnosis and treatment — https://doi.org/10.1186/s12903-023-03720-6
- See also: Study on remineralization of teeth with CPP-ACP and salivary pH analysis — https://doi.org/10.1038/s41405-023-00141-z
- See also: Randomized clinical trial on hydroxyapatite-containing toothpastes and caries-related variables — https://doi.org/10.1016/j.identj.2024.01.028

DOCUMENTS (2):
  • Study Protocol (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT07325643/Prot_000.pdf
  • Informed Consent Form (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT07325643/ICF_001.pdf